CLINICAL TRIAL: NCT01854775
Title: A Phase 2/3, Open-Label Study of the Pharmacokinetics, Safety, and Antiviral Activity of the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Single Tablet Regimen (STR) in HIV-1 Infected Antiretroviral Treatment-Naive Adolescents and Virologically Suppressed Children
Brief Title: Study to Evaluate the Pharmacokinetics, Safety, and Antiviral Activity of the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Single Tablet Regimen (STR) in HIV-1 Infected Antiretroviral Treatment-Naive Adolescents and Virologically Suppressed Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-0106; 2013-002780-26 (EudraCT Number)
Record Dates: First submitted 2013-05-03; First posted 2013-05-16 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Acquired Immune Deficiency Syndrome (AIDS); HIV Infections
Keywords: Adolescents; HIV-1; HIV; Treatment-naive; Virologically suppressed; Children
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg (Experimental): Treatment naive adolescents (12 to < 18 years of age) living with human immunodeficiency virus (HIV) will receive E/C/F/TAF (150/150/200/10 mg) fixed-dose combination (FDC) once daily for 48 weeks. Participants who complete 48 weeks of study treatment will have the option to receive E/C/F/TAF in an extension phase of the study until: a) the participant turns 18 years old and E/C/F/TAF is commercially available for adults in the country in which the participant is enrolled; b) age-appropriate E/C/F/TAF become commercially available in the country in which the participant is enrolled; or c) Gilead elects to terminate development of E/C/F/TAF in that country.
  Interventions: Drug: E/C/F/TAF
- Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg (Experimental): Children (6 to < 12 years of age weighing ≥ 25 kg) with HIV who were virologically suppressed will receive E/C/F/TAF (150/150/200/10 mg) FDC once daily for 48 weeks. Participants who complete 48 weeks of study treatment will have the option to receive E/C/F/TAF in an extension phase of the study until: a) the participant turns 18 years old and E/C/F/TAF is commercially available for adults in the country in which the participant is enrolled; b) age-appropriate E/C/F/TAF become commercially available in the country in which the participant is enrolled; or c) Gilead elects to terminate development of E/C/F/TAF in that country.
  Interventions: Drug: E/C/F/TAF
- Cohort 3: Age ≥2 Years and Weight ≥ 14 to <25 kg (Experimental): Children (≥ 2 years of age weighing ≥ 14 to < 25 kg) with HIV who were virologically suppressed will receive E/C/F/TAF (90/90/120/6 mg) FDC once daily for 48 weeks. Participants who attain a weight of ≥ 25 kg during the course of the study will switch to adult E/C/F/TAF (150/150/200/10 mg) tablets administered orally, once daily with food. Participants who complete 48 weeks of study treatment will have the option to receive E/C/F/TAF in an extension phase of the study until: a) the participant turns 18 years old and E/C/F/TAF is commercially available for adults in the country in which the participant is enrolled; b) age-appropriate E/C/F/TAF became commercially available in the country in which the participant is enrolled; or c) Gilead elects to terminate development of E/C/F/TAF in that country.
  Interventions: Drug: E/C/F/TAF; Drug: E/C/F/TAF (Low Dose)

INTERVENTIONS:
Drug: E/C/F/TAF — Tablets administered orally with food.
  Other Names: Genvoya®
Drug: E/C/F/TAF (Low Dose) — 90/90/120/6 mg STR administered once daily orally with food.
  Arms: Cohort 3: Age ≥2 Years and Weight ≥ 14 to <25 kg

SUMMARY:
The primary objectives of Cohort 1 are to evaluate the steady state pharmacokinetics (PK) for elvitegravir (EVG) and tenofovir alafenamide (TAF) and confirm the dose of the elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) STR (Part A) and to evaluate the safety and tolerability of E/C/F/TAF STR through Week 24 (Part B) in human immunodeficiency virus - 1 (HIV-1) infected, antiretroviral (ARV) treatment-naive adolescents.

The primary objectives of Cohort 2 are to evaluate the PK of EVG and TAF (Part A), and to evaluate the safety and tolerability of E/C/F/TAF through Week 24 (Part B) in virologically suppressed HIV-1 infection children 6 to < 12 years weighing >= 25 kg.

The primary objectives of Cohort 3 are to evaluate the PK of EVG and TAF and confirm the dose of the STR, and to evaluate the safety and tolerability of E/C/F/TAF low dose (LD) STR in virologically suppressed HIV-1 infected children ≥ 2 years of age and weighing ≥ 14 to < 25 kg.

ELIGIBILITY:
Key Inclusion Criteria:

* Cohort 1

  * Age at baseline: 12 years to < 18 years old
  * Weight at screening: ≥ 35 kg (77 lbs)
  * Plasma HIV-1 ribonucleic acid (RNA) levels of ≥ 1,000 copies/mL at screening (Roche COBAS TaqMan v2.0)
  * Screening genotype report shows sensitivity to EVG, emtricitabine (FTC) and tenofovir (TFV)
  * No prior use of any approved or experimental anti-HIV-1 drug for any length of time
* Cohort 2

  * Age at baseline: 6 years to < 12 years old
  * Weight at screening: ≥ 25 kg (55 lbs)
  * Plasma HIV-1 RNA of < 50 copies/mL (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is > 50 copies/mL) for ≥ 180 consecutive days (6 months) prior to screening on a stable antiretroviral regimen, without documented history of resistance to any component of E/C/F/TAF STR.
* Cohort 3

  * Age at baseline: ≥ 2 years old
  * Weight at screening: ≥ 14 kg (31 lbs) to < 25 kg (55 lbs)
  * Plasma HIV-1 RNA: < 50 copies/mL (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is > 50 copies/mL) for ≥ 180 consecutive days (6 months) prior to screening on a stable antiretroviral regimen, without prior history of resistance to any component of E/C/F/TAF STR

Key Exclusion Criteria:

* Hepatitis B or hepatitis C virus infection
* Evidence of active pulmonary or extra-pulmonary tuberculosis disease within 3 months of the screening visit.
* Individuals experiencing decompensated cirrhosis
* Pregnant or lactating females

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2025-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- United States (5):
  - Miller's Children Hospital, Long Beach, California
  - Children's Research Institute, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington
- South Africa (6):
  - KIDCRU Ward J8, Cape Town
  - Be Part Yoluntu Centre, Cape Town
  - Desmond Tutu HIV Foundation, Cape Town
  - Perinatal HIV Research Unit Baragwanath Hospital, Johannesburg
  - Clinical HIV Research Unit, Johannesburg
  - Empilweni Services and Research Unit (ESRU), Johannesburg
- Thailand (3):
  - The HIV Netherlands Australia Thailand Research collaboration (HIV-NAT), Bangkok
  - Queen Savang Vadhana Memorial Hospital, Chon Buri
  - Department of Pediatrics, Faculty of Medicine, Khon Kaen University, Khon Kaen
- Joint Clinical Research Centre, Kampala, Uganda
- University of Zimbabwe - Clinical Research Centre, Belgravia, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Result] Rakhmanina N, Gaur A, Natukunda E, Chokephaibulkit K, Liberty A, Kido A, et al. Acceptability and palatability of the single-tablet regimens of B/F/TAF and E/C/F/TAF in children (6-12 years) living with HIV infection [Abstract 33]. 10th International Workshop on HIV Pediatrics; 2018 July 21-22; Amsterdam, The Netherlands
- [Result] Sharma S, Gupta S, Majeed S, Strehlau R, Hellstrom E, Liu Y, et al. Exposure-Safety of Tenofovir in Pediatric HIV-Infected Participants: Comparison of Tenofovir Alafenamide & Tenofovir Disoproxil Fumarate [Abstract 23]. 10th International Workshop on HIV Pediatrics; 2018 July 21-22; Amsterdam, The Netherlands.
- [Result] Natukunda E, Gaur AH, Kosalaraksa P, Batra J, Rakhmanina N, Porter D, Shao Y, Zhang H, Pikora C, Rhee MS. Safety, efficacy, and pharmacokinetics of single-tablet elvitegravir, cobicistat, emtricitabine, and tenofovir alafenamide in virologically suppressed, HIV-infected children: a single-arm, open-label trial. Lancet Child Adolesc Health. 2017 Sep;1(1):27-34. doi: 10.1016/S2352-4642(17)30009-3. Epub 2017 Jun 29. PMID 30169223
- [Result] Rakhmanina N, Natukunda E, Kosalaraksa P, Batra J, Gaur A, Shao Y, et al. Safety and efficacy of E/C/F/TAF in virologically suppressed, HIV-infected children through 48 weeks [Abstract 32]. 9th International Workshop on HIV Pediatrics; 2017 July 21-22; Paris, France.
- [Result] Gaur A, Natukunda E, Kosalarksa P, Batra J, Rakhmanina N, Coluci A, et al. Pharmacokinetics, Safety, and Efficacy of E/C/F/TAF in HIV-1-Infected Children (6 to <12 years) [Poster 424]. Conference on Retroviruses and Opportunistic Infections (CROI); 2017 February 13-16; Seattle Washington.
- [Result] Gaur AH, Kizito H, Prasitsueubsai W, Rakhmanina N, Rassool M, Chakraborty R, Batra J, Kosalaraksa P, Luesomboon W, Porter D, Shao Y, Myers M, Ting L, SenGupta D, Quirk E, Rhee MS. Safety, efficacy, and pharmacokinetics of a single-tablet regimen containing elvitegravir, cobicistat, emtricitabine, and tenofovir alafenamide in treatment-naive, HIV-infected adolescents: a single-arm, open-label trial. Lancet HIV. 2016 Dec;3(12):e561-e568. doi: 10.1016/S2352-3018(16)30121-7. Epub 2016 Oct 17. PMID 27765666
- [Result] Gaur A, Kizito H, Chakraborty R, Batra J, Kosalaraksa P, Luesomboon W, et al. Safety and Efficacy of E/C/F/TAF in HIV-1 Infected Treatment-Naive Adolescents [Poster 817]. Conference on Retroviruses and Opportunistic Infections (CROI); 2016 February 22-25; Boston, Massachusetts.
- [Result] Natukunda E, Liberty A, Strehlau R, Hellstrom E, Hakim JG, Kaur H, et al. Safety, pharmacokinetics and efficacy of low dose E/C/F/TAF in virologically suppressed children ≥ 2 years old living with HIV. (Abstract OABLB0101) 23rd International AIDS Conference; 06-10 July 2020 (Virtual).
- [Result] Natukunda E, Liberty A, Strehlau R, Hellstrom E, Hakim J, Kaur H, et al. Safety, pharmacokinetics, and efficacy of low dose E/C/F/TAF in virologically suppressed children ≥ 2 years old living with HIV. (Abstract 3) International Workshop on HIV Pediatrics 2020; 16-17 November 2020 (Virtual).
- [Result] Liberty A, Strehlau R, Rakhmanina N, Chokephaibulkit K, Koziara J, Kaur H, et al. Acceptability and palatability of low dose B/F/TAF and E/C/F/TAF in children (≥ 2y) with HIV. (Abstract 57) International Workshop on HIV Pediatrics 2020; 16-17 November 2020 (Virtual).
- [Result] Kizito H, Gaur A, Prasitsuebsai W, Rakhmanina N, Lawson E, Shao Y, et al. Safety, Efficacy and Pharmacokinetics of the Integrase Inhibitor-Based E/C/F/TAF Single-Tablet Regimen in Treatment-Naïve HIV-Infected Adolescents Through 24 Weeks of Treatment [Poster 953]. Conference on Retroviruses and Opportunistic Infections; 2015 February 23-26; Seattle, WA.
- [Result] Porter DP, Bennett SR, Quirk E, Miller MD, White KL. Lack of Emergent Resistance in HIV-1-Infected Adolescents on Elvitegravir-Based STRs [Poster 952]. Conference on Retroviruses and Opportunistic Infections (CROI); 2015 23-26 February; Seattle, WA.
- [Result] Kizito H, Gaur A, Prasitsuebsai W, Rakhmanina N, Lawson E, Shao Y, et al. Safety, Efficacy and Pharmacokinetics of the Integrase Inhibitor-Based E/C/F/TAF Single-Tablet Regimen in Treatment-Naïve HIV-Infected Adolescents Through 24 Weeks of Treatment [Poster 36]. 16th International Workshop on Clinical Pharmacology of HIV & Hepatitis Therapy; 2015 26-28 May; Washington, DC.
- [Result] Kizito H, Gaur A, Prasitsuebsai W, Rakhmanina N, Chokephaibulkit K, Fourie J, et al. Changes in renal laboratory markers and bone mineral density in treatment-naïve HIV-1-infected adolescents initiating INSTI-based single-tablet regimens containing tenofovir alafenamide (TAF) or tenofovir disoproxil fumarate (TDF) [Presentation #MOAB0104]. International AIDS Society (IAS) Conference on HIV Pathogenesis, Treatment and Prevention; 2015 19-22 July; Vancouver, Canada.
- [Result] Natukunda E, Gaur AH, Kosalaraksa P, Hellstrom E, Strehlau R, Liberty A, Cox S, Leisegang R, Palaparthy R, Crowe S, Vieira V, Kersey K, Rakhmanina N. Pharmacokinetics, safety and efficacy of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide in children with HIV aged from 2 years and weighing at least 14 kg. J Int AIDS Soc. 2025 Feb;28(2):e26414. doi: 10.1002/jia2.26414. PMID 39888251
- [Result] Natukunda E, Gaur AH, Deville JG, Kosalaraksa P, Strehlau R, Castano E, Liberty A, Crowe S, Palaparthy R, Vieira VA, Kersey K, Rakhmanina N, Gordon CM. Longitudinal Evaluation of Bone Safety in Children and Adolescents With HIV-1 Starting Tenofovir Alafenamide-Containing Antiretroviral Therapy. J Pediatric Infect Dis Soc. 2025 Aug 7;14(7):piaf062. doi: 10.1093/jpids/piaf062. PMID 40632108
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-292-0106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in South Africa, Thailand, Uganda, United States of America, and Zimbabwe.
Pre-assignment Details: 155 participants were screened.
Groups:
- Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg: Treatment naive adolescents (12 to < 18 years of age) with human immunodeficiency virus (HIV) received elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablets, once daily orally with food for 48 weeks. Participants who completed 48 weeks of study treatment had the option to receive E/C/F/TAF in an extension phase of the study until: a) the participant turned 18 years old and E/C/F/TAF was commercially available for adults in the country in which the participant was enrolled; b) age-appropriate E/C/F/TAF became commercially available in participant's country.
- Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg: Children (6 to < 12 years of age weighing ≥ 25 kg) with HIV who were virologically suppressed received E/C/F/TAF (150/150/200/10 mg) FDC tablets, once daily orally with food for 48 weeks. Participants who completed 48 weeks of study treatment had the option to receive E/C/F/TAF in an extension phase of the study until: a) the participant turned 18 years old and E/C/F/TAF was commercially available for adults in the country in which the participant was enrolled; b) age-appropriate E/C/F/TAF became commercially available in participant's country.
- Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg: Children (≥ 2 years of age weighing ≥ 14 to < 25 kg) with HIV who were virologically suppressed received E/C/F/TAF (90/90/120/6 mg) FDC tablets, once daily orally with food for 48 weeks. Participants who attained a weight of ≥ 25 kg during the course of the study were switched to adult E/C/F/TAF (150/150/200/10 mg) tablets administered orally, once daily with food. Participants who completed 48 weeks of study treatment had the option to receive E/C/F/TAF in an extension phase of the study until: a) the participant turned 18 years old and E/C/F/TAF was commercially available for adults in the country in which the participant was enrolled; b) age-appropriate E/C/F/TAF became commercially available in participant's country.
Period: Treatment Phase (48 Weeks)
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Started | 50 | 52 | 27
Completed | 48 | 51 | 27
Not Completed | 2 | 1 | 0
Not completed — Withdrew consent | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Extension Phase
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Started | 48 | 50 | 27
Completed | 44 | 49 | 27
Not Completed | 4 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Investigator's Discretion | 1 | 0 | 0
Not completed — Non-Compliance with study drug | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrew consent | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg | Total
Number analyzed (Participants) | 50 | 52 | 27 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.9) | 10 (1.2) | 6 (1.9) | 11 (3.7)
Age, Customized [Count of Participants; unit: Participants]
  2 to <6 Years | 0 | 0 | 11 | 11
  6 to <12 Years | 0 | 52 | 16 | 68
  12 to <18 Years | 50 | 0 | 0 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 17 | 75
  Male | 22 | 22 | 10 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 52 | 27 | 129
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 13 | 3 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 44 | 37 | 24 | 105
  White | 0 | 2 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 3 | 0 | 13 | 16
  Thailand | 6 | 13 | 1 | 20
  Uganda | 30 | 27 | 8 | 65
  United States | 11 | 12 | 3 | 26
  Zimbabwe | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Elvitegravir (EVG) (Cohort 1)
Description: AUCtau is defined as concentration of drug over time (the area under the concentration versus time curve over the dosing interval).
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 5 minutes, 0.25, 0.5, 1, 1.5, 2, 4, 5, 8 and 24 hours post-dose at Week 4
Population: The PK Substudy Analysis Set included all enrolled and treated participants from Part A who had any nonmissing key PK parameters (AUCtau, AUClast, Cmax) from Week 4 intensive PK data for the respective analyte.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 24
hr*ng/mL | 23840.1 (6076.15)

2. Primary Outcome: PK Parameter: AUCtau of EVG (Cohort 2)
Description: as for outcome 1
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 22
hr*ng/mL | 33813.9 (19536.30)

3. Primary Outcome: PK Parameter: AUCtau of EVG (Cohort 3)
Description: as for outcome 1
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, and 8 hours post-dose at Week 2
Population: The Intensive PK Analysis Set included all enrolled and treated participants who had any nonmissing key PK parameters (AUCtau, AUClast, Cmax) from Week 2 intensive PK data for the respective analyte.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 24
hr*ng/mL | 33245.6 (15499.22)

4. Primary Outcome: PK Parameter: AUClast of Tenofovir Alafenamide (TAF) (Cohort 1)
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration, area under the concentration time curve to last observation (AUClast).
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 5 minutes, 0.25, 0.5, 1, 1.5, 2, 4, 5, 8 and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 24
hr*ng/mL | 188.9 (105.45)

5. Primary Outcome: PK Parameter: AUClast of TAF (Cohort 2)
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 23
hr*ng/mL | 332.9 (149.12)

6. Primary Outcome: PK Parameter: AUCtau of TAF (Cohort 3)
Description: as for outcome 1
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, and 8 hours post-dose at Week 2
Population: Participants in the Intensive PK Analysis Set (all enrolled and treated participants who had any nonmissing key PK parameters [AUCtau, AUClast, Cmax] from Week 2 intensive PK data for the respective analyte) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 17
hr*ng/mL | 366.4 (144.91)

7. Primary Outcome: Cohort 1: Percentage of Participants With All Treatment-Emergent Adverse Events (AEs) and Treatment-Emergent Serious Adverse Events (SAEs)
Description: Treatment-emergent adverse events (TEAEs) were defined as any AEs that begin or worsen on or after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the Gilead Sciences Grading Scale for Severity of Adverse Events. An AE that met one or more of the following outcomes was classified as serious:
  * Fatal
  * Life-threatening
  * Disabling/incapacitating
  * Results in hospitalization or prolongs a hospital stay
  * A congenital abnormality
  * Other important medical events may also be considered serious AEs if they may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From first dose date up to Week 24
Population: Participants in the Safety Analysis Set (all participants who received at least 1 dose of study drug) with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 48
percentage of participants
  Any TEAEs | 81.3
  SAEs | 8.3

8. Primary Outcome: Cohort 2: Percentage of Participants With All Treatment-Emergent AEs and Treatment-Emergent SAEs
Description: TEAEs were defined as any AEs that begin or worsen on or after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the Gilead Sciences Grading Scale for Severity of Adverse Events. An AE that met one or more of the following outcomes was classified as serious:
  * Fatal
  * Life-threatening
  * Disabling/incapacitating
  * Results in hospitalization or prolongs a hospital stay
  * A congenital abnormality
  * Other important medical events may also be considered serious AEs if they may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From first dose date up to Week 24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 23
percentage of participants
  Any TEAEs | 73.9
  SAEs | 0

9. Primary Outcome: Cohort 3: Percentage of Participants With All Treatment-Emergent AEs and Treatment-Emergent SAEs
Description: as for outcome 8
Time Frame: From first dose date up to Week 24
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of participants
  Any TEAEs | 70.4
  SAEs | 3.7

10. Secondary Outcome: PK Parameter: Ctau of EVG, Emtricitabine (FTC), Tenofovir (TFV), and Cobicistat (COBI) (Cohort 1)
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 5 minutes, 0.25, 0.5, 1, 1.5, 2, 4, 5, 8 and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 24
ng/mL
  EVG | 300.8 (243.69)
  FTC: number analyzed (Participants) | 23
  FTC | 102.4 (39.85)
  TFV | 10.0 (2.13)
  COBI: number analyzed (Participants) | 15
  COBI | 25.0 (44.97)

11. Secondary Outcome: PK Parameter: Ctau of EVG, FTC, TFV and COBI (Cohort 2)
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 23
ng/mL
  EVG | 370.0 (438.52)
  FTC | 114.9 (27.70)
  TFV | 15.1 (3.77)
  COBI | 96.0 (162.01)

12. Secondary Outcome: PK Parameter: Ctau of EVG, FTC, TFV, and COBI (Cohort 3)
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, and 8 hours post-dose at Week 2
Population: Participants in the Intensive PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
ng/mL
  EVG: number analyzed (Participants) | 22
  EVG | 277.5 (223.43)
  FTC | 82.5 (26.47)
  TFV | 11.4 (2.65)
  COBI: number analyzed (Participants) | 18
  COBI | 23.0 (23.02)

13. Secondary Outcome: PK Parameter: Cmax of EVG, TAF, FTC, TFV, and COBI (Cohort 1)
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 5 minutes, 0.25, 0.5, 1, 1.5, 2, 4, 5, 8 and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 24
ng/mL
  EVG | 2229.6 (427.93)
  TAF | 166.8 (107.44)
  FTC | 2265.0 (510.55)
  TFV | 17.6 (4.18)
  COBI | 1202.4 (421.21)

14. Secondary Outcome: PK Parameter: Cmax of EVG, TAF, FTC, TFV, and COBI (Cohort 2)
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 23
ng/mL
  EVG | 3055.2 (1180.90)
  TAF | 313.3 (191.68)
  FTC | 3397.4 (916.06)
  TFV | 26.1 (5.43)
  COBI | 2079.4 (970.81)

15. Secondary Outcome: PK Parameter: Cmax of EVG, TAF, FTC, TFV, and COBI (Cohort 3)
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, and 8 hours post-dose at Week 2
Population: Participants in the Intensive PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
ng/mL
  EVG | 3297.2 (1720.38)
  TAF | 286.6 (206.97)
  FTC | 3007.4 (1138.10)
  TFV | 19.6 (4.72)
  COBI | 1525.5 (788.12)

16. Secondary Outcome: PK Parameter: CL/F of EVG and TAF (Cohort 1)
Description: Apparent oral clearance (CL/F) is defined as the apparent clearance of the drug following oral administration.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 5 minutes, 0.25, 0.5, 1, 1.5, 2, 4, 5, 8 and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 24
L/hr
  EVG | 6.7 (1.74)
  TAF: number analyzed (Participants) | 23
  TAF | 68.6 (52.64)

17. Secondary Outcome: PK Parameter: CL/F of EVG and TAF (Cohort 2)
Description: CL/F is defined as the apparent clearance of the drug following oral administration.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 22
L/hr
  EVG | 6.3 (5.11)
  TAF: number analyzed (Participants) | 11
  TAF | 31.9 (11.21)

18. Secondary Outcome: PK Parameter: CL/F of EVG and TAF (Cohort 3)
Description: CL/F is defined as the apparent clearance of the drug following oral administration.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, and 8 hours post-dose at Week 2
Population: Participants in the Intensive PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 24
L/hr
  EVG | 3.4 (1.79)
  TAF: number analyzed (Participants) | 17
  TAF | 18.5 (6.27)

19. Secondary Outcome: PK Parameter: Vz/F of EVG and TAF (Cohort 1)
Description: Vz/F is defined as the apparent volume of distribution of the drug after oral administration.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 5 minutes, 0.25, 0.5, 1, 1.5, 2, 4, 5, 8 and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 24
liters
  EVG | 60.5 (18.77)
  TAF: number analyzed (Participants) | 23
  TAF | 49.7 (32.54)

20. Secondary Outcome: PK Parameter: Vz/F of EVG and TAF (Cohort 2)
Description: Vz/F is defined as the apparent volume of distribution of the drug after oral administration.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 14
liters
  EVG | 46.8 (36.02)
  TAF: number analyzed (Participants) | 11
  TAF | 28.6 (25.74)

21. Secondary Outcome: PK Parameter: Vz/F of EVG and TAF (Cohort 3)
Description: Vz/F is defined as the apparent volume of distribution of the drug after oral administration.
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, and 8 hours post-dose at Week 2
Population: Participants in the Intensive PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 17
liters
  EVG: number analyzed (Participants) | 14
  EVG | 28.5 (28.30)
  TAF | 16.3 (11.07)

22. Secondary Outcome: PK Parameter: AUCtau of FTC, TFV, and COBI (Cohort 1)
Description: as for outcome 1
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 5 minutes, 0.25, 0.5, 1, 1.5, 2, 4, 5, 8 and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 24
hr*ng/mL
  FTC | 14424.4 (3452.88)
  TFV: number analyzed (Participants) | 23
  TFV | 287.6 (54.09)
  COBI: number analyzed (Participants) | 23
  COBI | 8240.8 (2972.94)

23. Secondary Outcome: PK Parameter: AUCtau of FTC, TFV, and COBI (Cohort 2)
Description: as for outcome 1
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose at Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 23
hr*ng/mL
  FTC: number analyzed (Participants) | 22
  FTC | 20629.2 (3906.01)
  TFV | 440.2 (92.13)
  COBI: number analyzed (Participants) | 20
  COBI | 15890.7 (8208.78)

24. Secondary Outcome: PK Parameter: AUCtau of FTC, TFV, and COBI (Cohort 3)
Description: as for outcome 1
Time Frame: 0 (pre-dose, ≤ 30 minutes prior to dosing), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, and 8 hours post-dose at Week 2
Population: Participants in the Intensive PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
hr*ng/mL
  FTC | 19468.1 (5635.74)
  TFV | 334.9 (76.77)
  COBI: number analyzed (Participants) | 21
  COBI | 14485.2 (7166.10)

25. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, as Defined by the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: The Full analysis set included all participants who were enrolled in the study and had received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of participants | 90.0

26. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, as Defined by the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of participants | 92.0

27. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 24, as Defined by the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 400 Copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of participants | 94.0

28. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 48, as Defined by the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 400 Copies/mL at Weeks 24 and 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of participants | 94.0

29. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, as Defined by the FDA Snapshot Analysis
Description: as for outcome 25
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0 [93.2 to 100.0]

30. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, as Defined by the FDA Snapshot Analysis
Description: as for outcome 26
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 98.1 [89.7 to 100.0]

31. Secondary Outcome: Cohort 3: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, as Defined by the FDA Snapshot Analysis
Description: as for outcome 25
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of participants | 96.3 [81.0 to 99.9]

32. Secondary Outcome: Cohort 3: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, as Defined by the FDA Snapshot Analysis
Description: as for outcome 26
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of participants | 96.3 [81.0 to 99.9]

33. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, Based on Missing = Failure Analyses
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed based on missing = failure analyses.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of participants | 90.0 [78.2 to 96.7]

34. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, Based on Missing = Failure Analyses
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed based on missing = failure analyses.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of participants | 92.0 [80.8 to 97.8]

35. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 24, Based on Missing = Failure Analyses
Description: as for outcome 33
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of participants | 94.0

36. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 48, Based on Missing = Failure Analyses
Description: The percentage of participants with HIV-1 RNA < 400 copies/mL at Week 48 was analyzed based on missing = failure analyses.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of participants | 94.0

37. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, Based on Missing = Failure Analyses
Description: as for outcome 33
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0 [93.2 to 100.0]

38. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, Based on Missing = Failure Analyses
Description: as for outcome 34
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0 [93.2 to 100.0]

39. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 24, Based on Missing = Failure Analyses
Description: The percentage of participants with HIV-1 RNA < 400 copies/mL at Week 24 was analyzed based on missing = failure analyses.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0

40. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 48, Based on Missing = Failure Analyses
Description: as for outcome 36
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0

41. Secondary Outcome: Cohort 3: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, Based on Missing = Failure Analyses
Description: as for outcome 33
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of participants | 96.3 [81.0 to 99.9]

42. Secondary Outcome: Cohort 3: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, Based on Missing = Failure Analyses
Description: as for outcome 34
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of participants | 96.3 [81.0 to 99.9]

43. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, Based on Missing = Excluded Analyses
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed based on missing = excluded analyses.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 48
percentage of participants | 93.8 [82.8 to 98.7]

44. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, Based on Missing = Excluded Analyses
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed based on missing = excluded analyses.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 48
percentage of participants | 95.8 [85.7 to 99.5]

45. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 24, Based on Missing = Excluded Analyses
Description: The percentage of participants with HIV-1 RNA < 400 copies/mL at Week 24 was analyzed based on missing = excluded analyses.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 48
percentage of participants | 97.9

46. Secondary Outcome: Cohort 1: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 48, Based on Missing = Excluded Analyses
Description: The percentage of participants with HIV-1 RNA < 400 copies/mL at Week 48 was analyzed based on missing = excluded analyses.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 48
percentage of participants | 97.9

47. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, Based on Missing = Excluded Analyses
Description: as for outcome 43
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0 [93.2 to 100.0]

48. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, Based on Missing = Excluded Analyses
Description: as for outcome 44
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0 [93.2 to 100.0]

49. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 24, Based on Missing = Excluded Analyses
Description: as for outcome 45
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0

50. Secondary Outcome: Cohort 2: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 48, Based on Missing = Excluded Analyses
Description: as for outcome 46
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of participants | 100.0

51. Secondary Outcome: Cohort 3: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 24, Based on Missing = Excluded Analyses
Description: as for outcome 43
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of participants | 96.3 [81.0 to 99.9]

52. Secondary Outcome: Cohort 3: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 48, Based on Missing = Excluded Analyses
Description: as for outcome 44
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of participants | 96.3 [81.0 to 99.9]

53. Secondary Outcome: Cohort 1: Change From Baseline in Plasma log10 HIV-1 RNA at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
copies/mL
  Baseline | 4.62 (0.587)
  Change at Week 24: number analyzed (Participants) | 48
  Change at Week 24 | -3.25 (0.645)

54. Secondary Outcome: Cohort 1: Change From Baseline in Plasma log10 HIV-1 RNA at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
copies/mL
  Baseline | 4.62 (0.587)
  Change at Week 48: number analyzed (Participants) | 48
  Change at Week 48 | -3.26 (0.712)

55. Secondary Outcome: Cohort 1: Change From Baseline in Cluster of Differentiation (CD4+) Cell Count at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
cells/μL
  Baseline | 471 (212.2)
  Change at Week 24: number analyzed (Participants) | 48
  Change at Week 24 | 191 (175.2)

56. Secondary Outcome: Cohort 1: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
cells/μL
  Baseline | 471 (212.2)
  Change at Week 48: number analyzed (Participants) | 47
  Change at Week 48 | 224 (170.3)

57. Secondary Outcome: Cohort 2: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
cells/μL
  Baseline | 961 (275.5)
  Change at Week 24 | -118 (194.1)

58. Secondary Outcome: Cohort 2: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
cells/µL
  Baseline | 961 (275.5)
  Change at Week 48: number analyzed (Participants) | 50
  Change at Week 48 | -66 (203.6)

59. Secondary Outcome: Cohort 3: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
cells/μL
  Baseline | 1153 (459.9)
  Change at Week 24: number analyzed (Participants) | 17
  Change at Week 24 | -137 (278.3)

60. Secondary Outcome: Cohort 3: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
cells/µL
  Baseline | 1153 (459.9)
  Change at Week 48: number analyzed (Participants) | 24
  Change at Week 48 | -179 (319.2)

61. Secondary Outcome: Cohort 1: Change From Baseline in CD4+ Cell Percentage at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ cell
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of CD4+ cell
  Baseline | 23.6 (8.80)
  Change at Week 24: number analyzed (Participants) | 48
  Change at Week 24 | 7.7 (4.77)

62. Secondary Outcome: Cohort 1: Change From Baseline in CD4+ Cell Percentage at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ cell
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg
Number analyzed (Participants) | 50
percentage of CD4+ cell
  Baseline | 23.6 (8.80)
  Change at Week 48: number analyzed (Participants) | 47
  Change at Week 48 | 9.3 (5.19)

63. Secondary Outcome: Cohort 2: Change From Baseline in CD4+ Cell Percentage at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ cell
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of CD4+ cell
  Baseline | 38.2 (6.44)
  Change at Week 24 | -0.8 (3.97)

64. Secondary Outcome: Cohort 2: Change From Baseline in CD4+ Cell Percentage at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ cell
Arm/Group | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg
Number analyzed (Participants) | 52
percentage of CD4+ cell
  Baseline | 38.2 (6.44)
  Change at Week 48: number analyzed (Participants) | 50
  Change at Week 48 | -0.6 (4.37)

65. Secondary Outcome: Cohort 3: Change From Baseline in CD4+ Cell Percentage at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ cell
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of CD4+ cell
  Baseline | 35.9 (6.73)
  Change at Week 24: number analyzed (Participants) | 17
  Change at Week 24 | 0.0 (4.40)

66. Secondary Outcome: Cohort 3: Change From Baseline in CD4+ Cell Percentage at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ cell
Arm/Group | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
Number analyzed (Participants) | 27
percentage of CD4+ cell
  Baseline | 35.9 (6.73)
  Change at Week 48: number analyzed (Participants) | 24
  Change at Week 48 | 0.2 (3.78)

ADVERSE EVENTS:
Time Frame: Up to 583 Weeks
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/52 | 0/27
Serious Adverse Events (participants affected / at risk) | 10/50 | 7/52 | 1/27
Other Adverse Events (participants affected / at risk) | 47/50 | 45/52 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg (N=50) | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg (N=52) | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg (N=27)
Uveitis (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Abortion infected (Infections and infestations) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Sinusitis bacterial (Infections and infestations) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Behaviour disorder (Psychiatric disorders) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 0
Glomerulonephritis acute (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Age 12 to < 18 Years and Weight ≥ 35 kg (N=50) | Cohort 2: Age 6 to < 12 Years and Weight ≥ 25 kg (N=52) | Cohort 3: Age ≥ 2 Years and Weight ≥ 14 to < 25 kg (N=27)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 | 3 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0 | 1
Visual impairment (Eye disorders) | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 10 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 4 | 3
Dental caries (Gastrointestinal disorders) | 7 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 14 | 7 | 2
Gastritis (Gastrointestinal disorders) | 7 | 2 | 0
Nausea (Gastrointestinal disorders) | 15 | 2 | 0
Vomiting (Gastrointestinal disorders) | 12 | 13 | 4
Pyrexia (General disorders) | 3 | 3 | 2
Anal gonococcal infection (Infections and infestations) | 3 | 0 | 0
Body tinea (Infections and infestations) | 7 | 0 | 2
Bronchitis (Infections and infestations) | 2 | 2 | 2
Conjunctivitis (Infections and infestations) | 4 | 1 | 0
Covid-19 (Infections and infestations) | 2 | 3 | 1
Folliculitis (Infections and infestations) | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 3 | 1
Hordeolum (Infections and infestations) | 3 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Malaria (Infections and infestations) | 14 | 4 | 0
Nasal herpes (Infections and infestations) | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 5
Oral herpes (Infections and infestations) | 3 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 2
Otitis media acute (Infections and infestations) | 2 | 0 | 2
Pharyngitis (Infections and infestations) | 4 | 0 | 3
Pneumonia (Infections and infestations) | 6 | 1 | 1
Respiratory tract infection (Infections and infestations) | 19 | 11 | 4
Rhinitis (Infections and infestations) | 3 | 0 | 1
Tinea capitis (Infections and infestations) | 2 | 4 | 2
Tonsillitis (Infections and infestations) | 6 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 20 | 14 | 14
Urinary tract infection (Infections and infestations) | 9 | 5 | 3
Vulvovaginal candidiasis (Infections and infestations) | 5 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 3 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Weight decreased (Investigations) | 4 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 8 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 1
Dizziness (Nervous system disorders) | 6 | 2 | 0
Headache (Nervous system disorders) | 14 | 8 | 1
Somnolence (Nervous system disorders) | 3 | 0 | 0
Product size issue (Product Issues) | 5 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 2
Heavy menstrual bleeding (Reproductive system and breast disorders) | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 0
Acne (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 7 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Study Protocol: Protocol Amendment 6 (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT01854775/Prot_000.pdf
  • Study Protocol: Protocol Amendment 7 (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT01854775/Prot_003.pdf
  • Statistical Analysis Plan: Interim 4 Analysis (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT01854775/SAP_001.pdf
  • Statistical Analysis Plan: Interim 6 Analysis (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT01854775/SAP_002.pdf
  • Statistical Analysis Plan: Final Analysis (2025-08-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT01854775/SAP_004.pdf